CLINICAL TRIAL: NCT02191293
Title: Long-term Observational Study in Patients Under Anti-retroviral Combination Therapy Who Were Switched From Protease Inhibitors or Other NNRTI to Viramune® Plus Two Nucleoside Reverse Transcriptase Inhibitors (NRTI) for Reasons of Therapy. (Long-Term Switch)
Brief Title: Long-term Study in Patients Under Anti-retroviral Combination Therapy Switching to Viramune®
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1402
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Viramune®
  Interventions: Drug: Viramune® tablets

INTERVENTIONS:
Drug: Viramune® tablets

SUMMARY:
Collecting data on maintaining anti-retroviral activity (quantitative HIV RNA determination) and immunological activity (CD4 cells) after switching from protease inhibitor or NNRTI to Nevirapine (Viramune®) and collecting of routinely observed laboratory data on lipids, and liver enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female out-patients with HIV type 1 infection who have achieved a viral load below detection limit (50 copies/ml) for more than 6 months under a previous combination therapy with protease-inhibitors (PI) or non-nucleoside reverse transcriptase inhibitors (NNRTI)
* Women can only be included, if a test has excluded pregnancy
* Only women can be included, who use a reliable means of contraception during the observational study

Exclusion Criteria:

* Known sensitivity to Viramune or one of its excipients
* Clinically relevant changes in lab findings (e.g. increase in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) by more than five-fold of upper limit normal)
* Patient is not able to abstain from treatment with ketoconazole, oral contraceptives, and other medication CYP3A metabolism
* For females:

  * Pregnancy
  * Breast-feeding
  * Insufficient or unreliable contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV treatment centres and HIV out-patient facilities
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2002-05; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Changes in viral load (HIV-RNA) | Baseline, up to 36 months
Changes in CD4 cell count | Baseline, up to 36 months

SECONDARY OUTCOMES:
Changes in body weight | Baseline, up to 36 months
Changes in general well-being assessed on a 4-point scale | Baseline, up to 36 months
Changes in lipid parameters | Baseline, up to 36 months
  mg/dl
Changes in glucose | Baseline, up to 36 months
  mg/dl
Changes in liver enzymes | Baseline, up to 36 months
  U/l
Number of patients with adverse events | up to 36 months